CLINICAL TRIAL: NCT00570323
Title: A Phase II Trial of Neoadjuvant Arimidex With or Without Faslodex in Postmenopausal Women With Hormone Receptor Positive Breast Cancer
Brief Title: Arimidex With or Without Faslodex In Postmenopausal Women With HR Positive Breast Cancer
Acronym: PACT001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mothaffar Rimawi (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Mothaffar Rimawi, Medical Director, Baylor Breast Care Center
Organization: Baylor Breast Care Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H 20431; IRUSFULV0060 (Other: AstraZeneca)
Record Dates: First submitted 2007-12-06; First posted 2007-12-10 (Estimated); Results first posted 2019-03-04 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; HORMONE RECEPTOR POSITIVE BREAST CANCER
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ARM A / Arimidex with Faslodex (Active Comparator): Arimidex with Faslodex in postmenopausal women
  Interventions: Drug: Arimidex; Drug: Faslodex
- ARM B Arimidex without Faslodex (Active Comparator): Arimidex without Faslodex in postmenopausal women.
  Interventions: Drug: Arimidex

INTERVENTIONS:
Drug: Arimidex — Aromatase inhibitors
  Other Names: Anastrozole
Drug: Faslodex — Hormone Receptor
  Other Names: Fulvestrant
  Arms: ARM A / Arimidex with Faslodex

SUMMARY:
Over the last 3 decades, a steady shift has occurred in the management of breast cancer. Because it was traditionally viewed as a local disease, many advocated the use of radical surgery to achieve maximum survival benefit. This view has been slowly replaced by a broader biologic view that recognizes the often systemic nature of breast cancer, even when it appears to be localized to the breast. Results from randomized clinical trials have demonstrated that less extensive surgery, or lumpectomy plus radiation therapy, are optimal for local management of early breast cancer. In addition to the less radical approach to surgical treatment of breast cancer, other randomized clinical trials have established the value of postoperative systemic therapy in improving overall survival by eradicating micrometastatic disease, the major cause of mortality from breast cancer. Despite the well-documented benefits of adjuvant systemic therapy, it is not effective in preventing death from breast cancer in all patients who are candidates for such treatment. The worth of such therapy can only be judged in retrospect upon disease relapse, a time when breast cancer is nearly always incurable. Currently, there are few reliable methods to predict the success or failure of a particular postoperative treatment modality, and better ways to predict and optimize outcome are needed.

Combination endocrine therapy: Using endocrine agents with different mechanisms of action together has the potential advantage of more effectively blocking ER signaling, thus improving the efficacy of such agents against breast cancer. In the past, attempts to combine endocrine agents for ER-positive breast cancer have had mixed results, depending on the setting and the patient population studied.

Endocrine agents without any agonist effect could potentially be used in combination with aromatase inhibitors, under the rationale that the combination would maximally blockade estrogen receptor signaling, thus potentially improving the antitumor effect. Fulvestrant (FASLODEX) is a pure estrogen antagonist with no known agonist effect; thus, it has the potential to provide additional benefit when combined with an aromatase inhibitor. This concept provides the rationale for using the combination of anastrazole and fulvestrant in this study.

DETAILED DESCRIPTION:
Purpose and Objectives

The primary objective of this study is to determine if ER-targeted therapy, ARIMIDEX and FASLODEX, used in combination is superior to ARMIDEX alone in hormone receptor positive breast cancer.

Primary study objective 1. To determine the efficacy of primary breast cancer, as measured by decrease in proliferation (KI67), to the combination of ARIMIDEX, and FASLODEX at high dose

Secondary study objectives 1. To study molecular changes in response to treatment. 2. To correlate changes in Ki67 with clinical response 3. To determine the pathologic response rate. 4. To assess the tolerability and safety of the combination regimen.

This is a phase II randomized multi-center study. As indicated in the study design schema found in the protocol document attached to Section S, patients will be initially randomized to receive ARIMIDEX, or ARIMIDEX+FASLODEX (high dose) for 16 weeks (112 days). A computer-generated randomization scheme will be generated by the study statistician at the Breast Center, Baylor College of Medicine. A 1:1 randomization scheme using permuted blocks will be employed. Randomization will be centralized at the Breast Center, Baylor College of Medicine and accomplished via access to a secure web-based procedure that is currently being implemented in our other multi-center clinical trials. Enrollment, eligibility, and randomization information will be stored in an Oracle database on the Breast Center's Sun server and will be accessible only through secure web-based applications. Communication with the pharmacy will be handled by email which will contain only patient identification number and initials and by FAX or hardcopy. The hardcopy will be used by physicians to send to the pharmacy a signed computer-generated pharmacy order to legally dispense study drug.

Within 30 days prior to randomization subjects will sign the study consent form, and have a history and physical exam, including all concurrent medications. Blood will be drawn for CBC, platelets, serum chemistries, BUN, creatinine, and liver function tests. If necessary to determine menopausal status FSH, LH and serum estradiol will be obtained. An EKG, CXR PA and lateral will be performed and a bilateral mammogram and US of primary breast cancer will be done within 90 days of randomization. Subjects will then be randomized to receive either ARIMIDEX 1 mg po q day (Group A), or ARIMIDEX 1 mg po q day and FASLODEX 500 mg IM, day 1, day 14, day 28 and thereafter once every 28 days (Group B). Study medications will be dispensed within 60 days of randomization. On day 28, subjects will be evaluated for side effects and a second breast core biopsy will be obtained. Evaluation for tumor response and tolerability of the regimen will be evaluated every 28 days in outpatient clinic visits. ALL treatment will continue until day 112 when patients with a clinical response or stable disease will receive appropriate surgical resection. If the tumor is unresectable on day 112, a core needle biopsy will be done. The surgical specimen will be obtained for further molecular analysis. After surgery, patients will be off study and will receive additional breast cancer therapy at the discretion of their treating physician. Patients who develop progressive disease on protocol will be taken off study and offered alternative treatment. All patients will have a safety follow-up 1 month after the surgery (or the alternative core biopsy).

Treatment will be administered on outpatient basis. After the baseline breast biopsy, patients will be randomized to receive ARIMIDEX 1mg po q day (group A), or ARIMIDEX 1mg po q day with FASLODEX 500 mg day 1, day 14, day 28, and thereafter every 28 days (Group B). After 28 days a second biopsy will be obtained in all patients. All patients will continue on the same randomized treatment for the total duration of the study of 112 days till the day before surgery. No investigational or commercial agents or therapies other than those described below may be administered with the intent to treat the patient's malignancy.

Study Visit Procedures: Pre-Study Procedures will include the following: informed consent, breast biopsy, demographics, medical history, concurrent medication list, physical exam, blood draw, bidimensional tumor measurement, bilateral mammogram, primary breast ultrasound and chest x-ray.

Day 1 procedures will include the following: study drug administration, clinic visit.

Day 14 procedures will include the following (group B only) study drug injection and clinic visit.

Day 28 procedures will include the following (group B only) study drug injection. Both group A and B, breast biopsy, concurrent medication list, physical exam, blood draw, clinic visit, adverse events evaluation, bidimensional tumor measurement.

Day 56 procedures will include the following (group B only) study drug injection. Both group A and B, concurrent medication list, physical exam, blood draw, adverse events evaluation, clinic visit and bidimensional tumor measurement.

Day 84 procedures include (group B only) study drug injection. Both group A and B, concurrent medication list, physical exam, blood draw, adverse event evaluation, clinic visit and bidimensional tumor measurement.

Day 112 procedures include study drug administration, concurrent medication list, physical exam, blood draw, adverse events evaluation, bidimensional tumor measurement, bilateral mammogram, primary breast ultrasound and tumor resection.

Day 140 procedures include blood draw, clinic visit and safety evaluation for adverse events.

Duration of Therapy In the absence of treatment delays due to adverse events, treatment will continue for 4 months or until one of the following criteria applies: Disease progression, Intercurrent illness that prevents further administration of treatment, Unacceptable adverse events(s), Patient decides to withdraw from the study, or General or specific changes in the patient's condition render the patient unacceptable for further treatment in the judgment of the investigator.

This protocol will close 6 months after the last patient is enrolled. Patients will receive study medications from day 0 until day 111, which is the day before their planned surgery. On day 140, patients will have a safety follow up visit and to determine the need for further treatment after surgery.

Breast Core Biopsy All subjects will have a breast tumor core biopsy at the beginning of the study, and a second biopsy after 2 weeks. Core needle biopsies are planned because they will provide sufficient histologically evaluable tissue for the assays proposed in this study.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must be female.
* Postmenopausal status, defined as any one of the following criteria:

  * Documented history of bilateral oophorectomy.
  * Age 60 years or more.
  * Age 45 to 59 and satisfying one or more of the following criteria:

    * Amenorrhea for at least 12 months and intact uterus.
    * Amenorrhea for less than 12 months and a follicle stimulating hormone (FSH) and estradiol concentration within postmenopausal range including: patients who have had a hysterectomy and patients who have received hormone replacement.
* Patients must have histologically confirmed invasive breast cancer with a primary tumor of 3 cm or more in greatest dimension as measured by clinical examination.
* Estrogen receptor and/or progesterone receptor positive disease.
* Patients must not have received any prior treatment for current or newly diagnosed breast cancer.
* Patients must have not received previous treatment with any of the study medications or similar drugs.
* No use of selective estrogen receptor modulators (SERM) such as raloxifene or similar agents in the past 2 years.
* WHO performance status of 0, 1, or 2.
* Adequate organ function defined as follows:

  * Adequate renal function, defined by a serum creatinine within 3 times the upper limits of normal.
  * Adequate liver function, defined by total bilirubin, AST, ALT, and alkaline phosphatase within 3 times the upper limits of normal.
  * Adequate bone marrow function, defined as a WBC greater than 3.0 ml, PLT greater than 75,000/ul, Hb greater than 9 gm/l.
* Willing to undergo breast core biopsies as required by the study protocol. - Ability to understand and sign a written informed consent for participation in the trial.
* Life expectancy of at least 1 year.

Exclusion Criteria:

* Premenopausal status.
* Other coexisting malignancies with the exception of basal cell carcinoma or cervical cancer in situ.
* Patients with brain metastasis.
* WHO performance status of 3 or 4.
* Is judged by the investigator, uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, significant cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the subject to participate in the clinical trial. - Concurrent treatment with estrogens or progestins. Patients must stop these drugs at least two weeks prior to study entry.
* Treatment with a non-approved or investigational drug within 30 days before Day 1 of study treatment.
* Platelet count less than 75,000.
* In the opinion of the investigator, bleeding diathesis or anticoagulation therapy that would preclude intramuscular injections.
* History of hypersensitivity to castor oil.
* Any evidence of clinically active interstitial lung disease (patients with chronic stable radiographic changes who are asymptomatic need not be excluded) - Patients with recurrent breast cancer.
* Patients with contralateral second primary breast cancers are eligible.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2007-12 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2018-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mothaffar Rimawi, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arimidex With Faslodex: Arimidex with Faslodex in postmenopausal women
  Arimidex with Faslodex: Arimidex with Faslodex
- Arimidex: Arimidex without Faslodex in postmenopausal women.
  Arimidex without Faslodex: Arimidex without Faslodex
Period: Started Treatment After Randomization
Arm/Group | Arimidex With Faslodex | Arimidex
Started | 36 | 36
Completed | 34 | 35
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Physician Decision | 1 | 0
Period: Complete Study After Start
Arm/Group | Arimidex With Faslodex | Arimidex
Started | 34 | 35
Completed | 31 | 34
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arimidex With Faslodex | Arimidex | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Continuous [Median (Full Range); unit: years] | 63 [51 to 87] | 59 [49 to 76] | 61 [49 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 36 | 72
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 11 | 26
  Not Hispanic or Latino | 21 | 25 | 46
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 10 | 17
  White | 28 | 23 | 51
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Ki-67 Levels From Baseline (Pre) to Day 28 (Post) Biopsy Samples
Description: The primary endpoint is change in Ki-67 levels from baseline (pre) to day 28 (post) biopsy samples. Ki-67 levels were log-transformed to achieve approximately normally distributed data. The differences in these log-transformed values between post vs. pre biopsy samples were calculated. This difference represents the log of the ratio of post vs. pre Ki-67 levels in the original scale.
Time Frame: baseline (pre) to day 28 (post)
Population: Patients were evaluable if their baseline and day28 samples were collected and the samples werer in good quality. 30 patients were excluded from the analysis: 12 patients did not provide the samples at baseline and/or day28; another 18 patients' samples were found with no tumor.
Measure: Mean (Standard Deviation); unit: log-transformed Ki67%
Arm/Group | ARM A / Arimidex With Faslodex | ARM B Arimidex Without Faslodex
Number analyzed (Participants) | 22 | 20
log-transformed Ki67% | -1.3632 (0.8949) | -1.6237 (2.1592)
Statistical Analysis 1: Comparison: ARM A / Arimidex With Faslodex vs ARM B Arimidex Without Faslodex; Test type: Superiority; p = 0.6202, t-test, 2 sided

2. Secondary Outcome: Clinical Response
Description: Measurable lesions were examined at baseline to treatment completion.Clinical Response was defined by Solid Tumor Response Criteria (RECIST).
Time Frame: 1 Year
Population: Patients who completed the study treatment were evaluable. 7 patients who did not complete the treatment were excluded from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arimidex With Faslodex | Arimidex
Number analyzed (Participants) | 31 | 34
Participants
  Complete response | 4 | 5
  Partial response | 18 | 19
  Stable disease | 5 | 5
  Progression disease | 4 | 5

3. Secondary Outcome: Pathologic Complete Response
Description: Pathologic response was defined as no residual invasive tumor on histopathological analysis in the breast primary. Patients were assessed according to the Chevallier classification of pathologic response.
Time Frame: 1 Year
Population: Patients who had surgery in the study were evaluable. 13 patients who did not have surgery were excluded from the analysis: 7 patients did not complete study treatment, another 6 patients did not have surgery performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Arimidex With Faslodex | Arimidex
Number analyzed (Participants) | 29 | 30
Participants
  pathologic response | 1 | 2
  not pathologic response | 28 | 28

ADVERSE EVENTS:
Arm/Group | Arimidex | Arimidex With Faslodex
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/34
Other Adverse Events (participants affected / at risk) | 25/35 | 22/34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arimidex (N=35) | Arimidex With Faslodex (N=34)
Arthralgia (Nervous system disorders) | 13 (14) | 7 (7)
Bone pain (Nervous system disorders) | 4 (4) | 3 (3)
Fatigue (General disorders) | 8 (9) | 7 (7)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Headache (Nervous system disorders) | 3 (4) | 3 (3)
Hot flashes (Endocrine disorders) | 16 (16) | 11 (11)
Insomnia (General disorders) | 6 (6) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 5 (5)
Vaginal dryness (Reproductive system and breast disorders) | 6 (6) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes